CLINICAL TRIAL: NCT06518902
Title: A Single Arm, Open Label Exploratory Clinical Study on the Safety, Tolerability, and Preliminary Efficacy of Mesenchymal Stem Cells (Umbilical Cord) Injection in the Treatment of Acute Ischemic Stroke (AIS) Patients
Brief Title: Umbilical Cord-derived Mesenchymal Stem Cell Infusion for Treating Acute Ischemic Stroke
Acronym: UMERIS
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Engineering Center of Cell Products (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSCTAISP-01
Record Dates: First submitted 2024-07-18; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSCs group (Experimental): mesenchymal stem cells (umbilical cord) injection once or once a week for three consecutive weeks.
  Interventions: Drug: mesenchymal stem cells (umbilical cord) injection

INTERVENTIONS:
Drug: mesenchymal stem cells (umbilical cord) injection — Patients receive mesenchymal stem cells (umbilical cord) injection once or once a week for three consecutive weeks

SUMMARY:
The goal of this clinical trial is to learn if drug mesenchymal stem cells (umbilical cord) injection works to treat acute ischemic stroke in adults. It will also learn about the safety and efficacy of drug mesenchymal stem cells (umbilical cord) injection . The main questions it aims to answer are:

Identify the dose-limiting toxicity (DLT) of drug mesenchymal stem cells (umbilical cord) injection in acute ischemic stroke patients.

Dose the drug mesenchymal stem cells (umbilical cord) injection improves the mRS score, NIHSS score, Fugl-Meyer score and and Barthel index of acute ischemic stroke patients? What is the pharmacokinetic characteristics and immunogenic response of mesenchymal stem cells (umbilical cord) injection in the treatment of acute ischemic stroke patients.

What is the the possible molecular mechanisms of mesenchymal stem cells (umbilical cord) injection in the treatment of acute ischemic stroke patients.

Participants will:

Take drug drug mesenchymal stem cells (umbilical cord) injection once or once a week for three consecutive weeks.

After receiving the corresponding dose of mesenchymal stem cells (umbilical cord) injection, the subjects entered a 6-month safety, efficacy observation and further safety evaluation period. Long term efficacy and survival follow-up up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age range of 18-80 years old (including threshold), gender not limited;
2. The clinical diagnosis of this episode is anterior circulation ischemic stroke, confirmed by MRI/CT, and the patient can receive experimental drugs within one month after the onset of stroke symptoms;
3. Individuals with a National Institutes of Health Stroke Scale (NIHSS) score of 6-20 (inclusive) and a NIHSS score of Ia<2 points;
4. Female subjects with fertility or male subjects with fertility partners who have no fertility plans and voluntarily take effective contraceptive measures during the study period;
5. Individuals with self-reported or family reported mRS scores of 0 or 1 prior to the onset of current stroke symptoms;
6. After receiving complete information about the study, all participants voluntarily participate in the clinical study by signing an informed consent form themselves or their guardians.

Exclusion Criteria:

1. Individuals with epilepsy, Alzheimer's disease, Parkinson's disease, severe depression, or other neurological disorders or mental illnesses that researchers believe may affect their ability to participate in trials or impact research evaluations;
2. Bleeding transformation occurred, and according to the researchers' judgment, it is not suitable to participate in clinical trials;
3. Patients with malignant tumors, excluding low-grade malignant tumors such as basal cell carcinoma, papillary thyroid carcinoma, and localized prostate cancer in situ, who have received curative treatment for more than five years;
4. Serious infections, including sepsis, septic shock, severe pneumonia (diagnostic criteria for severe pneumonia refer to the 2007 American College of Infectious Diseases/American Thoracic Society diagnostic criteria for adult severe pneumonia), etc;
5. Patients with respiratory failure, or those with current evidence of pulmonary embolism or suspected pulmonary embolism;
6. Organ function levels that meet any one or more of the following criteria:

   1. ALT or AST>2 × ULN; TBil>1.5×ULN； Scr>2×ULN；
   2. Thrombocytopenia (platelet count<75000/mm3) or heparin induced thrombocytopenia;
   3. For patients who have not received anticoagulant therapy, activated partial thromboplastin time (APTT)>2.5 × ULN or prothrombin time (PT)>2.5 × ULN; Patients who have received anticoagulant therapy and have been assessed by researchers to have a serious risk of bleeding;
   4. Hemoglobin (Hb)<90g/L;
7. Individuals who have had or currently have severe cardiovascular disease:

   1. Suffering from CTCAE grade II or above myocardial ischemia or myocardial infarction, or unstable angina pectoris;
   2. Researchers believe that severe arrhythmias with clinical significance;
   3. NYHA standard III-IV cardiac dysfunction;
   4. Other acute and severe complications that endanger life;
8. Poorly controlled hypertensive patients (defined as those who have undergone antihypertensive treatment but have sustained systolic blood pressure>220mmHg or diastolic blood pressure>120mmHg);
9. Poorly controlled diabetes (defined as blood glucose still>16.8 mmol/L after treatment) or hypoglycemia (blood glucose<2.8 mmol/L);
10. Individuals with a history of immunodeficiency, including HIV positive, other acquired or congenital immunodeficiency diseases, idiopathic IgA deficiency, or those who require systemic steroid hormone (≥ 10 mg/day of prednisone equivalent)/immunosuppressive drug treatment within 14 days prior to or during the trial period;
11. Patients who are positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb), as well as positive for HBV DNA, hepatitis C antibody (HCV), or Treponema pallidum antibody (TPAb/PRR);
12. Screening individuals who have participated in clinical trials of other drugs within the previous 3 months;
13. Individuals known to be allergic to the investigational drug or any component of the investigational drug (including human serum albumin, dimethyl sulfoxide, or compound electrolyte injection, as well as bovine derived products);
14. Individuals who are unable to undergo cranial CT/MRI examination due to various reasons;
15. Patients who have undergone major surgery, suffered severe trauma, or plan to undergo neurological function assessment during the trial period within the 3 months prior to the first administration of medication;
16. Breastfeeding or pregnant women (pregnancy diagnosis is evaluated through a combination of blood pregnancy test/urine pregnancy test and/or obstetric ultrasound examination);
17. Combining other serious systemic diseases, or having a medical history of any disease or laboratory abnormality that may confuse the study results, interfere with subject participation in the study procedure, or not be in the best interest of subject participation in the study, based on the researcher's judgment, is not suitable for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 6 months
  Dose-limiting toxicity and Maximum tolerated dose

IPD SHARING:
Plan to Share IPD: Undecided